CLINICAL TRIAL: NCT00094991
Title: Mechanism of Action and Efficacy of Muraglitazar (BMS298585) in the Treatment of Type 2 Diabetic Patients
Brief Title: Mechanism of Action and Efficacy of Muraglitazar in Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV168-026
Record Dates: First submitted 2004-10-29; First posted 2004-11-01 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2007-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — muraglitazar

INTERVENTIONS:
Drug: Muraglitazar

SUMMARY:
The purpose of this study is to learn more about how muraglitazar lowers blood sugar in people with type 2 diabetes. The safety of this treatment will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes;
* Serum triglyceride concentration < or = 600 mg/dL;
* Body mass index < or = 37 kg/m2

Exclusion Criteria:

* Type 1 diabetes;
* History of myocardial infarction (MI), coronary angioplasty, bypass graft(s), valvular disease, unstable angina pectoris, transient ischemic attack (TIA), or cerebrovascular accident (CVA) within 6 months;
* Congestive heart failure (NYHA Class III and IV);
* Uncontrolled hypertension;
* Women of Child Bearing Potential
* History of renal disease, peripheral vascular disease (PVD), pulmonary disease, gastrointestinal disease, active liver disease, or endocrine disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42
Dates: Start 2004-05; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
The change from baseline in insulin medicated glucose disposal after 16 weeks of treatment with Muraglitazar

CONTACTS AND LOCATIONS:
Locations (2):
- Local Institution, San Antonio, Texas, United States
- Local Institution, Pisa, Italy